CLINICAL TRIAL: NCT05274529
Title: Effects of Personal Technology Driven Workplace Wellbeing Intervention Programme on Wellbeing, Productivity (Presenteeism) and Absenteeism - an Intervention Study
Acronym: Coachbeat
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Firstbeat Technologies Oy (Industry)
Collaborators: Aisti Health Oy (Unknown); University of Jyvaskyla (Other); Tampere University (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: Coachbeat
Record Dates: First submitted 2022-01-26; First posted 2022-03-10 (Actual); Last update posted 2024-03-05 (Actual); Status verified 2024-03

CONDITIONS: Occupational Stress; Occupational Burnout
Keywords: workplace; wellbeing; intervention; absenteeism; presenteeism; stress; burnout
MeSH Terms: conditions — Occupational Stress; Burnout, Professional; Burnout, Psychological | interventions — Mental Health; Pliability; Sleep; Salvage Therapy

STUDY DESIGN:
Intervention Model Description: This is a pre-post type intervention study where baseline measurements are made at 0 months from the study start and follow up measurements are made at 4, 8 ,12, 24 and 36 months.
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Study group (Experimental): All the participants will be in the same group and have the same intervention programmes options to choose from.
  Interventions: Behavioral: Psychological health and flexibility; Behavioral: Work ability; Behavioral: Sleep and recovery; Behavioral: Healthy lifestyle; Other: No coaching

INTERVENTIONS:
Behavioral: Psychological health and flexibility — A remote coaching programme concentrating on psychological health and flexibility
Behavioral: Work ability — A remote coaching programme concentrating on work ability
Behavioral: Sleep and recovery — A remote coaching programme concentrating on sleep and recovery
Behavioral: Healthy lifestyle — A remote coaching programme concentrating on healthy lifestyle
Other: No coaching — Participants also have the option to choose no coaching for the coming 3 month period.

SUMMARY:
In this study the effects of a technology-driven workplace wellbeing intervention programme on employees' wellbeing, productivity (presenteeism) and absenteeism will be studied with the help of mobile applications and remotely conducted questionnaires, different wellbeing intervention periods and HRV based measurements.

DETAILED DESCRIPTION:
The objectives of this study are:

1. To study the effects of a data driven adaptive workplace wellbeing intervention programme on productivity (presenteeism) and absenteeism of the employees.
2. To study the effects of data driven adaptive workplace wellbeing interventions on employees' physical health measures and wellbeing. The secondary objective also includes studying whether the programme generates measurable financial savings.

This study is an intervention study where eligible participants will be offered a technologically delivered health promotion intervention which is personalized to their needs both in terms of content and timing within the 12-month intervention period. The outcomes are compared against their pre-intervention levels at both individual and group level. The study has no control group as it is not acceptable for the participating companies to offer participation only to part of their employees based on randomization due to expected positive impact of the intervention. The lack of the control group will be taken into account while analyzing and interpreting the study results.

The 12-month intervention period consists of access to Firstbeat Life (HRV & movement measurement based wellbeing service), Aava Medical's Aisti wellbeing assessment and four types of online coaching programmes plus option of no coaching. Every participant has continuous access to Firstbeat Life and Aisti during the entire intervention programme and may use them at any time they so desire. In addition, participants will use the Coachbeat mobile app which is used to instruct and communicate with the participants, to fill in all the study questionnaires at given times, and to promote use of Firstbeat Life and Aisti at given points of the study. Baseline measurements and measurements after 4 and 8 months give recommendations for participation to the online coaching based on Firstbeat Life and Aisti wellbeing assessment. The participants can choose the coaching program based on the recommendation or their own interest. They can participate several coaching programmes during the study. Each coaching programme lasts approximately 3 months.

ELIGIBILITY:
The initial target population consists of generally healthy employees of selected employer companies from information intensive industries and jobs.

Inclusion Criteria:

* Signed written informed consent
* Adequate Finnish or English1 language skills to comprehend study-related instructions and questionnaires. The services and contents are available only in Finnish and English.

Exclusion Criteria:

* Planned absenteeism from work during the study with >3mth duration
* Use of cardiac pacemaker or history of atrial fibrillation
* No access to compatible mobile phone
* History of a major cardiovascular event (myocardial infarction, coronary artery bypass graft (CABG), percutaneous coronary intervention (PCI), stroke, or transient ischemic attack) within the previous 6 months

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 571 (Actual)
Dates: Start 2022-04-12 (Actual); Primary Completion 2026-10 (Estimated); Study Completion 2026-10 (Estimated)

PRIMARY OUTCOMES:
The change in work productivity loss (presenteeism) by WLQ | 0, 4, 8, 12, 24 and 36 months from start
  The change in work productivity loss (presenteeism) is assessed by repeating Work Limitations Questionnaires (WLQ). WLQ results are on a scale from 0 to 100 where 0 means no limitations to work (=best result) and 100 means the most limitations to work (=worst result)
The change in work productivity loss (presenteeism) by HPQ | 0, 4, 8, 12, 24 and 36 months from start
  The change in work productivity loss (presenteeism) is assessed by repeating Health and Work Performance Questionnaires (HPQ). HPQ scale goes from 0 to 10 where 10 means the best health and work performance.
The change in work ability | 0, 12, 24 and 36 months from start
  The change in work ability is assessed by repeating work ability index (WAI) questionnaires. WAI scores are on a scale from 7 to 49 points where 7 is the poorest and 49 is the best work ability.
The change in sick-leaves (absenteeism) by absenteeism records | 0, 12, 24 and 36 months from start
  The change in sick-leaves (absenteeism) are assessed via employer absenteeism records
The change in sick-leaves (absenteeism) by HPQ | 0, 12, 24 and 36 months from start
  The change in sick-leaves (absenteeism) are assessed via repeating Health and Work Performance Questionnaires (HPQ). HPQ scale goes from 0 to 10 where 10 means the best health and work performance.
The change in sick-leaves (absenteeism) by WAI | 0, 12, 24 and 36 months from start
  The change in sick-leaves (absenteeism) are assessed via repeating work ability index (WAI) questionnaires. WAI scores are on a scale from 7 to 49 points where 7 is the poorest and 49 is the best work ability.

SECONDARY OUTCOMES:
The change in autonomic nervous system function and health behaviors based on HRV | 0, 4, 8, 12, 24 and 36 months from start
  The change in autonomic nervous system function and health behaviors is assessed by HRV (heart rate variability)
The change in autonomic nervous system function and health behaviors based on measured stress/recovery | 0, 4, 8, 12, 24 and 36 months from start
  The change in autonomic nervous system function and health behaviors is assessed by measured stress/recovery. Stress & recovery balance is scored on a scale from 0 to 100 in Firstbeat Life service (100 is the best score)
The change in autonomic nervous system function and health behaviors based on measured sleep | 0, 4, 8, 12, 24 and 36 months from start
  The change in autonomic nervous system function and health behaviors is assessed by measured sleep. Sleep is scored on a scale from 0 to 100 in Firstbeat Life service (100 is the best score)
The change in autonomic nervous system function and health behaviors based on measured physical activity | 0, 4, 8, 12, 24 and 36 months from start
  The change in autonomic nervous system function and health behaviors is assessed by measured physical activity. Physical activity is scored on a scale from 0 to 100 in Firstbeat Life service (100 is the best score)
The change in autonomic nervous system function and health behaviors based on measured physical fitness | 0, 4, 8, 12, 24 and 36 months from start
  The change in autonomic nervous system function and health behaviors is assessed by measured physical fitness as assessed by VO2Max
The change in depression and mood by BBI-15 | 0 and 12 months from start
  The change in depression and mood are assessed by Bergen Burnout Indicator (BBI-15). BBI-15 result is on a scale from 0 to 100 where scores from 0 to 74 mean "no burnout" and scores from 95 to 100 mean "severe burnout".
The change in self-reported questionnaire measures | 0, 12, 24 and 36 months from start
  Self-reported questionnaire measures are mental wellbeing, physical health, sleep and recovery, financial situation, social relationships, work-related information etc. in the Aisti Index wellbeing assessment. Aisti assessment gives results on a scale from 0 to 100 (100 is best) for each area of life.
The change in blood pressure | 0 and 12 months from start
  The change in blood pressure is measured between the start and the end of the 12 month intervention period.
The change in weight | 0 and 12 months from start
  The change in weight is measured between the start and the end of the 12 month intervention period.
The change in waist circumference | 0 and 12 months from start
  The change in waist circumference is measured between the start and the end of the 12 month intervention period.
The change in neck circumference | 0 and 12 months from start
  The change in neck circumference is measured between the start and the end of the 12 month intervention period.
Return of investment (ROI) | 0, 12, 24 and 36 months from start
  Return of investment (ROI) is calculated through absenteeism statistics and self-reported presenteeism.
Company's financial performance | 0, 12, 24 and 36 months from start
  Company's financial performance is evaluation is based on reported revenue and profit.

CONTACTS AND LOCATIONS:
Overall Officials: Jari Parkkari, Dr, Study Chair — Professor at University of Jyväskylä; Tero Myllymäki, M.Sc., Principal Investigator — Head of Physiology Research at Firstbeat Technologies
Locations (1):
- Aisti Health Oy, Helsinki, Finland